CLINICAL TRIAL: NCT07268937
Title: Assessment of Hepatic Steatosis Using Dedicated Software Implemented on Ultrasound Devices
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Gianluigi Poma, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: p_168
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CAP (Controlled Attenuation Parameter) module implemented on the Fibroscan machine. — Use of the CAP module implemented on the Fibroscan machine to compare the results of the degree of steatosis

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is currently the most common chronic liver disease, with an estimated prevalence of 5-30% in the general population and 55-80% in patients with type 2 diabetes.

Methods for the quantitative and non-invasive assessment of liver fat content have recently been implemented on ultrasound devices, based on the estimation of the ultrasound beam attenuation coefficient and backscattering. These methods are CE marked and already commercially available.

The aim of the study is to compare the results of the degree of steatosis detected by different ultrasound devices with the degree of steatosis of the CAP (Controlled Attenuation Parameter) module implemented on the Fibroscan machine.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* ability to hold breath for image acquisition,
* informed consent

Exclusion Criteria:

* withdrawal of informed consent,
* any condition which, in the clinical judgement of the investigator, will make further participation in the study unacceptable for that individual patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an age > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the results relating to the degree of steatosis detected by the various ultrasound devices with the CAP module | 05 May 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SSD Malattie Infettive 3 - Ecografia, Pavia, Pavia, Italy